CLINICAL TRIAL: NCT07102810
Title: Standardized Hypnotic Susceptibility Testing to Facilitate Development of a Machine Learning Tool to Characterize Physiological Biomarkers of Calm and Tranced States
Brief Title: Hypnosis-Based Machine Learning Biomarker Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: Entrancing Entertainment, Inc. (Unknown)
Responsible Party: Principal Investigator, David Reich, Professor of Anesthesiology, Perioperative and Pain Medicine, Icahn School of Medicine at Mount Sinai
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY-25-00767
Record Dates: First submitted 2025-07-30; First posted 2025-08-05 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Disorder; Trance; Anxiety
Keywords: Hypnosis; Trance; Anxiety; Machine Learning; Calm
MeSH Terms: conditions — Osteopetrosis, mild autosomal recessive form; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: This project will facilitate within-subjects and between-subjects comparisons in a limited number of subjects exposed to a standardized hypnotic susceptibility protocol -- the Harvard Group Scale of Hypnotic Susceptibility (HGSHS:A). This is a widely used test to assess an individual's susceptibility to hypnotic suggestion. The State Trait Anxiety Inventory (STAI) will be perform immediately prior to and following the hypnotic protocol. Together, these reliable and valid data will serve as the gold standards to facilitate training of a machine-learning model that will attempt to use physiological data (EEG and wearable-derived) and high-resolution audiovisual recordings of subject/hypnotist responses to develop a patient monitoring tool that measures emotional/arousal states spanning the spectrum from anxiety through calm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Guided Hypnosis (Experimental): All participants will undergo a single, standardized hypnotic susceptibility protocol using the Harvard Group Scale of Hypnotic Susceptibility: Form A (HGSHS:A).
  Interventions: Behavioral: Standardized Hypnotic Susceptibility Testing

INTERVENTIONS:
Behavioral: Standardized Hypnotic Susceptibility Testing — Participants will be guided through the Harvard Group Scale of Hypnotic Susceptibility: Form A (HGSHS:A), a validated group hypnosis protocol that includes standardized hypnotic inductions and suggestibility tasks.
  Other Names: HGSHS:A

SUMMARY:
This study seeks to contribute to the growing body of literature on hypnosis by providing robust, data-driven insights into the physiological mechanisms underlying trance states. The integration of electroencephalogram (EEG) and other wearable-derived physiological data will offer a comprehensive assessment of the changes that occur during a standardized hypnosis protocol: the Harvard Group Scale of Hypnotic Susceptibility (HGSHS:A). The results of this study are intended to facilitate derivation and validation of an Artificial Intelligence/Machine Learning (AI/ML)-based monitor that quantifies a patient's instantaneous emotional/arousal state along the spectrum that spans anxiety through states of calmness and trance. Future investigations will explore the ability of using such an interactive virtual system as a component of a closed-loop adaptive device to create optimal states of non-pharmacological sedation using personalized audiovisual content to allay anxiety and discomfort during medical procedures, such as percutaneous biopsies.

DETAILED DESCRIPTION:
This is an interventional study that will acquire data to characterize the time course of physiological biomarkers and audiovisual observations of depth of trance before, during and upon emergence from a standardized hypnotic susceptibility protocol. The subjects will also complete the State Trait Anxiety Inventory (STAI) immediately before and after the hypnosis protocol. The differences in the biomarker signals among subjects of different degrees of hypnotic susceptibility and different pre-post levels of state anxiety will facilitate between- and within-subjects comparisons that will be supplemented by computer vision analysis of subject responses. The full data set will be used to facilitate derivation and validation of a novel machine-learning monitoring tool to measure instantaneous emotional/arousal levels along a spectrum that spans anxiety through calmness and trance.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent obtained from participant and ability and willingness for participant to comply with the requirements of the study.
* Adults of all genders, ages 18-65
* Healthy volunteers
* English-speaking

Exclusion Criteria:

* Participating currently in experimental drug trials.
* Recent (<1 year) or current history of substance use disorder.
* Diabetes T1 or T2, major cardiovascular or respiratory diseases, major neurological diseases, or limited mobility
* Presence of a condition or abnormality that in the opinion of the investigator would compromise the safety of the patient or the quality of the data.
* Adults that cannot consent.
* Chronic use of psychoactive medications.
* Chronic use of antiepileptic medications.
* Active substance use disorder.
* Participants reporting significant phobias or anxiety disorders triggered by imagery or situations involving insects (specifically flies), enclosed spaces or elevators (claustrophobia), or heights (acrophobia).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2025-08-04 (Actual); Primary Completion 2025-09-09 (Actual); Study Completion 2025-09-09 (Actual)

PRIMARY OUTCOMES:
Harvard Group Scale of Hypnotic Susceptibility (HGSHS:A) Total Score | During hypnosis session (single study visit)
  Total score (0-12) reflecting responsiveness to hypnotic suggestion during standardized protocol. Higher scores suggest greater responsiveness to hypnotic suggestion.

SECONDARY OUTCOMES:
State-Trait Anxiety Inventory (STAI) Subscale Scores | Immediately Pre- and immediately post-hypnosis session (single study visit)
  The State-Trait Anxiety Inventory is a 40-item instrument divided into two subscales: state and trait anxiety. State Subscale range from 20-80, with higher score suggesting more anxiety at a particular moment in time. Trait Subscale range from 20-80, with higher score suggesting general anxiety feelings overall. These will not be summed therefore there will not be one total scale.
EEG Spectral Power | Immediately Pre-, During, and immediately post-hypnosis session (single study visit)
  Power values in EEG frequency bands collected across 21 electrodes during baseline, hypnotic induction, and post-session phases.
Heart Rate (HR) | Immediately Pre-, During, and immediately post-hypnosis session (single study visit)
  Mean heart rate (beats per minute) captured continuously using a wearable chest patch before, during, and after hypnosis session.
Heart Rate Variability (HRV) | Immediately Pre-, During, and immediately post-hypnosis session (single study visit)
  Time and frequency domain HRV metrics derived from wearable ECG data.
Respiratory Rate (RR) | Immediately Pre-, During, and immediately post-hypnosis session (single study visit)
  Mean respiratory rate (breaths per minute) obtained from a respiration belt and ECG-derived signals.
Electrodermal Activity (EDA) | Immediately Pre-, During, and immediately post-hypnosis session (single study visit)
  Skin conductance level and phasic response rate measured using BIOPAC sensors.
Pre-Ejection Period (PEP) | Immediately Pre-, During, and immediately post-hypnosis session (single study visit)
  Pre-ejection period (ms), a marker of sympathetic nervous system activity, measured via seismocardiogram from chest patch.
Respiratory Sinus Arrhythmia (RSA) | Immediately Pre-, During, and immediately post-hypnosis session (single study visit)
  RSA index (ms²), derived from heart rate and respiration synchrony during hypnotic protocol.

CONTACTS AND LOCATIONS:
Overall Officials: David L Reich, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai Hospital
Locations (1):
- Mount Sinai Hospital, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
Aggregate deidentified data and results will be shared. Individual participant video and EEG data will not be shared due to PHI concerns.

DOCUMENTS (1):
  • Informed Consent Form (2025-07-15): https://cdn.clinicaltrials.gov/large-docs/10/NCT07102810/ICF_000.pdf